CLINICAL TRIAL: NCT05301452
Title: Evaluation of Intravascular Irradiation of Blood in Children With Sleep Bruxism - Study Protocol for a Randomized Controlled Clinical Trial
Brief Title: Evaluation of Intravascular Irradiation of Blood in Children With Sleep Bruxism
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ILIBSleepBruxism
Record Dates: First submitted 2022-03-16; First posted 2022-03-29 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Sleep Bruxism; Sleep Bruxism, Childhood
MeSH Terms: conditions — Sleep Bruxism | interventions — Myofunctional Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants will not know whether they belong to the placebo group, or the active photobiomodulation group, seeing as the laser application will be simulated.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): This group will receive an application of placebo ILIB and an orofacial myofunctional therapy (MFT) exercise protocol.
  Interventions: Radiation: Placebo Intravascular Irradiation of Blood (ILIB); Procedure: Orofacial Myofunctional Therapy
- ILIB Group (Active Comparator): This group will receive an application of ILIB and an orofacial myofunctional therapy (MFT) exercise protocol.
  Interventions: Radiation: Intravascular Irradiation of Blood (ILIB); Procedure: Orofacial Myofunctional Therapy

INTERVENTIONS:
Radiation: Intravascular Irradiation of Blood (ILIB) — The laser treatment will be performed by a speech therapist and will have the following parameters: wavelength of 808 nm. It will be done twice a week for 8 weeks, in 20-minute sessions.
  Arms: ILIB Group
Radiation: Placebo Intravascular Irradiation of Blood (ILIB) — The photobiomodulation procedure will be simulated, but with the laser turned off. It will be done twice a week for 8 weeks, in 20-minute sessions.
  Arms: Control Group
Procedure: Orofacial Myofunctional Therapy — Myofunctional therapy will be performed by a speech therapist specialized in the area. It will consist of 1 weekly session, where the functions of breathing, chewing and swallowing will be evaluated and addressed.
  The following exercises will be indicated: nasal hygiene, inflated cheeks with the tip of the tongue on the palate, lingual sweep, tongue thrust against the palate, tongue touch on the last molars, chewing of soft solids and bolus assembly (20 minute therapy session).

SUMMARY:
Background: The objective of this study will be to evaluate the effect of Intravascular Irradiation of Blood (ILIB) combined with myofunctional exercises for sleep bruxism in pediatrics. Methods: This study will be a randomized controlled clinical trial. A triage of individuals between 4 and 17 years old with a diagnosis of sleep bruxism will be carried out at the clinic of the Catholic University of Uruguay, and in a private office referred by different private care centers. The selected participants will be evaluated before and after treatment by means of questionnaires on bruxism, sleep quality and nocturnal oxygen saturation measurement. For this, 46 patients with sleep bruxism will be recruited, who will be divided into 2 groups: control group (CG), which will undergo an application of placebo ILIB and an orofacial myofunctional therapy (MFT) exercise protocol; and na ILIB group, which will carry out an active application of ILIB and an exercise protocol, this being once a week for 8 weeks. The laser treatment (808 nm) will be performed twice a week for 8 weeks. The values will be tested for normality by the Kolmogorov-Smirnov test. For the comparison between the groups, T-test will be carried out, considering a level of significance of 0.5% (p<0.05). Discussion: Although local photobiomodulation (PBM), acupuncture PBM and physiotherapy have been studied in the treatment of bruxism, this is the first study to evaluate the effect of ILIB combined with myofunctional exercises for sleep bruxism in pediatrics.

ELIGIBILITY:
Inclusion Criteria:

* in the mixed dentition phase (permanent incisors and first molars erupted);
* adolescents with an established permanent dentition.

Exclusion Criteria:

* People with dental caries;
* Those taking medications, such as inflammatory agents, muscle relaxants, corticosteroids, anticonvulsants, and antidepressants;
* Those with chronic diseases that affect muscles or motor coordination, and those who do not cooperate during the evaluation will be excluded from the study;
* Children with cerebral palsy;
* Patients whose guardians do not sign the informed consent or the user does not sign the assent.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-06-20 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Oximetry | Baseline and 8 weeks of treatment.
  A portable pulse oximeter that includes Masimo SET® Measure-through Motion and Low Perfusion™ pulse oximetry under motion and low perfusion conditions will be used. Nocturnal oximetry will be performed prior to treatment and post treatment. The parents or guardians of the minor will be trained.

SECONDARY OUTCOMES:
Changes in Breathing | Baseline and 8 weeks of treatment.
  A clinical evaluation will be carried out by a speech therapist specialized in the area of Orofacial Motricity, to check for possible improvement in breathing. It is the respiratory characterization from the taking of air, which explains the anatomical and topographical situation of its entrance to the respiratory system (respiratory mode), to the thoracoabdominal movement zone that integrates inspiration and expiration. It is supported by the observation with the aid of a Glatzel's mirror to anatomically determine the upper airway status and its functional correlation.
Changes in Swallowing | Baseline and 8 weeks of treatment.
  A clinical evaluation will be carried out by a speech therapist specialized in the area of Orofacial Motricity, to check for possible improvement in swallowing. For this, the Payne's test, which assesses tongue posture both at rest and in function (swallowing), will be used. From instruments such as liquid fluorescein applied to the apex lingual and lateral borders, and Payne's lamp that verifies the vestige of the fluroscein, and therefore the conditions of support, thrust, position and/or obstruction of the tongue.
Changes in Chewing | Baseline and 8 weeks of treatment.
  A clinical evaluation will be carried out by a speech therapist specialized in the area of Orofacial Motricity, to check for possible improvement in chewing. For this, the gnatodynamometer, test that allows to measure the force of the occlusion, will be used.
Changes in Speech | Baseline and 8 weeks of treatment.
  A clinical evaluation will be carried out by a speech therapist specialized in the area of Orofacial Motricity, to check for possible improvement in speech. For this, the Glatzel test will be used to measure the degree of nasal patency and the functional symmetry of the upper airways both at rest and in function. Specifically in the functional evaluation, its usefulness is linked to the verification of the existence of nasality or hyponasality before vowels elicited by the patient.
Changes in the Presence of Bruxism | Baseline and 8 weeks of treatment.
  The bruxism questionnaire will be delivered to parents or guardians, which will be completed prior to treatment and afterwards. The questionnaire contains 4 questions regarding the perceived presence of bruxism, and 5 questions for the dentist to answer, based on a clinical observation. All questions have the options "yes" or "no". The more times the word "yes" is chosen, the greater the risk for bruxism is.
Changes in Sleep Quality | Baseline and 8 weeks of treatment.
  A Pediatric Sleep Quality Questionnaire will be delivered to parents or guardians, and it will be completed prior to treatment and afterwards. The questionnaire contains 44 questions regarding sleep quality. All questions have the options "yes" or "no". The more times the word "yes" is chosen, the worse is the sleep quality.

REFERENCES:
- [Derived] Viarengo NO, Goncalves MLL, Bruno LH, Fossati AL, Sertaje MRF, Santos EM, Sobral APT, Mesquita-Ferrari RA, Fernandes KPS, Horliana ACRT, Motta LJ, Bussadori SK. Evaluation of intravascular irradiation of blood in children with sleep bruxism: Study protocol for a randomized controlled clinical trial. Medicine (Baltimore). 2022 Nov 4;101(44):e31230. doi: 10.1097/MD.0000000000031230. PMID 36343030